CLINICAL TRIAL: NCT06646445
Title: Neoadjuvant Pembrolizumab With a Watch-and-wait Strategy for Patients With Mismatch Repair-deficient or Microsatellite Instability-high (dMMR/MSI-H) Localized Colon Cancer: a Randomized GERCOR G-109 PRODIGE 84 PREMICES Phase II Trial
Brief Title: Neoadjuvant Pembrolizumab With a Watch-and-wait Strategy for dMMR/MSI-H Localized Colon Cancer: PREMICES Study.
Acronym: PREMICES
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Fondation ARCAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREMICES G-109 PRODIGE 84
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Colon Cancer
Keywords: pembrolizumab; watch-and-wait; microsatellite instability; mismatch repair deficient
MeSH Terms: conditions — Colonic Neoplasms; Microsatellite Instability; Turcot syndrome | interventions — pembrolizumab; Surgical Procedures, Operative; Chemotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: Pembrolizumab plus a watch-and-wait approach (experimental arm) Standard strategy (surgical resection ±adjuvant chemotherapy (control arm) 1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm A (Pembrolizumab plus watch-and-wait approach) (Experimental): Pembrolizumab and Watch-and-wait (TAP-CT scan, colonoscopy with biopsies)
  Interventions: Drug: Pembrolizumab Injection [Keytruda]; Procedure: Watch-and-wait approach
- Arm B (Surgical resection ± adjuvant chemotherapy) (Active Comparator): Standard of care surgery ± adjuvant chemotherapy (5-fluorouracil/capecitabine ± oxaliplatin 3 months to 6 months)
  Interventions: Procedure: Surgery; Drug: Adjuvant chemotherapy

INTERVENTIONS:
Drug: Pembrolizumab Injection [Keytruda] — Pembrolizumab 200 mg via a 30-minute IV infusion q3w on Day 1 of each 21-day cycle; 8 cycles ± 9 additional cycles (17 cycles in total).
  Other Names: Keytruda
  Arms: Experimental Arm A (Pembrolizumab plus watch-and-wait approach)
Procedure: Watch-and-wait approach — Watch-and-wait strategy:
  * TAP-CT scan At months 3 and 6 during 8 cycles of treatment, at months 9 and 12, and during additional 9 cycles of treatment if performed, and every 3 months thereafter for up to 2 years,
  * Colonoscopy with biopsies at months 3, 6, 9, 12, and 24.
  Arms: Experimental Arm A (Pembrolizumab plus watch-and-wait approach)
Procedure: Surgery — Standard of care surgery performed with a maximal delay of 21 days (3 weeks) from randomization.
  Arms: Arm B (Surgical resection ± adjuvant chemotherapy)
Drug: Adjuvant chemotherapy — Adjuvant chemotherapy (5-fluorouracil/capecitabine ± oxaliplatin 3 months to 6 months) according to the current guidelines, at the investigator's discretion.
  Arms: Arm B (Surgical resection ± adjuvant chemotherapy)

SUMMARY:
The goal of this investigational, multicenter, open-label randomized, two-stage phase II study is to evaluate neoadjuvant pembrolizumab with a watch-and-wait approach in patients with localized deficient mismatch repair / high microsatellite instability (dMMR/MSI-H) colorectal cancer (CRC). The PREMICES trial is based on the hypothesis that non-operative management is effective for dMMR/MSI-H localized CRC when treated with neoadjuvant pembrolizumab.

Eligible patients will be randomized in a 1:1 ratio to receive either pembrolizumab with a watch-and-wait approach (experimental arm A) or the standard strategy of surgical resection ± adjuvant chemotherapy (arm B).

DETAILED DESCRIPTION:
dMMR/MSI-H is a key biomarker for predicting the success of immune checkpoint inhibitors in colorectal cancer (CRC). Pembrolizumab has shown improved outcomes for patients with metastatic CRC, becoming the new standard of care. Neoadjuvant immunotherapy has demonstrated high rates of complete pathological responses in both metastatic and localized CRC, with promising results in non-surgical approaches. Studies support using a "watch-and-wait" strategy after immunotherapy, potentially avoiding surgery. These findings are reshaping treatment strategies for dMMR/MSI-H CRC, particularly regarding organ preservation and non-operative management.

The PREMICES study evaluates the efficacy of neoadjuvant pembrolizumab combined with a watch-and-wait approach for treating localized dMMR/MSI-H CRC. It investigates non-operative management as a potential strategy for achieving a complete clinical response in dMMR/MSI-H localized CRC without the need for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent (IC),
2. Aged ≥18 years,
3. An Eastern Cooperative Oncology Group Performance status (ECOG PS) of 0 or 1,
4. Newly diagnosed, histologically confirmed colonic or upper third rectal adenocarcinoma, NB: material must be available from biopsy done during colonoscopy.
5. Radiological tumor assessment at screening performed within 21 days before inclusion according to RECIST v1.1 by chest, abdomen, and pelvis (TAP- CT) showing resectable localized disease (cT0-4 cN0-2 cM0) and no metastatic disease,
6. dMMR and/or MSI-high (MSI-H) tumor status as follows:

   * loss of expression of ≥1 MMR protein (MLH1, MSH2, MSH6, or PMS2) or a dimeric couple (MLH1 and PMS2 or MSH2 and MSH6) on immunohistochemistry (IHC; using hMLH1, hMSH2, hMSH6, hPMS2 antibodies),
   * And/or ≥ 3 instable markers by the pentaplex by polymerase chain reaction (PCR) (BAT-25, BAT-26, NR-21, NR-24, and NR-27),

   NB:
   * In case of two instable markers by PCR, it is required to present confirmation of the dMMR status by IHC or comparison of PCR test with matched normal tissue.
   * In case of loss of expression of only one MMR protein by IHC or any other IHC pattern, it is required to confirm MSI status using pentaplex PCR; Agreement of Sponsor on a dMMR/MSI status is mandatory to include the patient (the patient's file [an anonymized mail] must be send to Sponsor before inclusion). Approval/refusal email for inclusion of the patient will be sent by Sponsor within 24 hours of receipt of the Investigator email. In case of discrepancy between IHC and PCR, the final decision about the dMMR/MSI status will be taken by Sponsor or coordinating investigator,
7. Adequate hematological status, renal, and liver function obtained within 14 days prior to randomization of study treatment:

   1. absolute neutrophil count (ANC) ≥1.5 x 10^9/L; platelets ≥100 x 10^9/L; hemoglobin ≥9 g/dL,
   2. serum creatinine level <150 µM or clearance >50 ml/min (Modification of the Diet in Renal Disease [MDRD] or Cockcroft and Gault),
   3. serum bilirubin ≤1.5 × upper limit of normal (ULN), alkaline phosphatase <5 x ULN, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 2.5 x ULN,
8. International normalized ratio (INR), prothrombin time (PT), and activated partial thromboplastin time (aPTT) ≤1.5 × ULN, except for the patient on anticoagulant therapy who must have PT-INR-aPTT within therapeutic range is deemed appropriate by the Investigator,
9. Has no contraindications to administration of oxaliplatin, capecitabine, or 5-fluorouracil, according to their respective summaries of product characteristics (SmPCs),
10. Is able to undergo surgery and receive adjuvant treatment (chemotherapy) as part of standard care,
11. A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

    1. Is a woman of non-childbearing potential as defined: i/ ≥45 years of age and has not had menses for >1 year, ii/ amenorrhea for <2 years without a hysterectomy and oophorectomy and have a high follicle stimulating hormone (FSH) value in the postmenopausal range upon pre-study (screening) evaluation, iii/ post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound, MRI, or CT scan,
    2. Negative pregnancy blood test within 72 hours before the first dose of pembrolizumab, AND
    3. If woman of childbearing potential (WOCBP), female patient must be willing to use a highly effective form of contraception (Appendix 24.9) from screening throughout the study treatment and 4 months after the last dose of pembrolizumab,
12. Male patient is eligible to participate if he agrees to the following during the study treatment and for 4 months after the last dose of pembrolizumab:

    1. Refrain from donating sperm,
    2. Must use contraception/barrier as follows:

       * Agree to use a male condom when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant.
       * Agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person,
13. Primary tumor tissue samples (archival or fresh biopsy specimen) acquired during coloscopy together with images availability (mandatory), NB: The patient's agreement will be specifically requested for endoscopic images in the patient information note and informed consent for their use as clinical data that may be analyzed and presented in publications. These data will be used in the same manner as other personal data. The confidentiality of these data will be maintained,
14. Patient willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study,
15. Registeration in the National Health Care System (PUMa - Protection Universelle Maladie included).

Exclusion Criteria:

1. Tumor that is not readily resectable,
2. Bifocal colorectal adenocarcinoma,
3. Locally advanced middle or low rectal cancer (<10 cm from the anal verge on MRI, sagittal slide) staged as cT3/T4 and/or N+ and/or with predictive circumferential margin >2 mm on pretreatment MRI, NB: for rectal cancers, the margin of the tumor relative to the anal margin should be indicated on the endoscopy report,
4. Major surgical procedure within 4 weeks prior to the first dose of study treatment,
5. Pre-existing hemostatic disorder or medical condition requiring chronic anticoagulation that cannot be interrupted for the purpose of study specified tumor resection or endoscopic biopsies,
6. Metastases (stage IV disease),
7. Has history of uncontrolled or symptomatic cardiac disease,
8. Prior treatment with an anti-PD(L)1, anti-LAG-3, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, including prior therapy with anti-tumor vaccines or other immuno-stimulatory antitumor agents,
9. Prior malignancy active within the previous 3 years apart from: i/ locally curable cancers that have been apparently cured (e.g., squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast); ii/ Lynch syndrome-related non-CRC in complete remission for > 1 year,
10. Patient is human immunodeficiency virus (HIV)-positive with CD4+ cell count <600 cell/ml or detectable viral load,
11. Has complete or partial dihydropyrimidine dehydrogenase deficiency (uracilemia ≥16 ng/ml), In particular, the uracilemia level must be determined before patient inclusion. Patients with altered uracilemia will be excluded.
12. Patient has active hepatitis B virus (HBV, defined as having a positive hepatitis B surface antigen [HBsAg] test) or hepatitis C virus (HCV) prior to inclusion, NB: Patients with past HBV infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible. NB: Patients positive for HCV antibody are eligible only if PCR testing is negative for HCV RNA.
13. Impossibility of submitting to the medical follow-up of the study for geographical, social, or psychiatric illness.
14. Patient under a legal protection regime (guardianship, curatorship, judicial safeguard) or administrative decision or incapable of giving his/her consent,

    Non-eligible to immunotherapy:
15. Any history of autoimmune disease including, but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis, NB: History of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.

    NB: Controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
16. Prior (non-infectious) pneumonitis requiring systemic corticosteroid therapy or has currently pneumonitis,
17. Any live, attenuated vaccine within 30 days prior to the first dose of study treatment or such administration is anticipated during the study,
18. Prior allogeneic bone marrow transplantation or prior solid organ transplantation,
19. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 14 days (2 weeks) prior to the first dose of trial treatment or is required to receive systemic immunosuppressive medications during the study. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
20. Ongoing anti-cancer treatment for another cancer (to be discussed with the coordinator in case of hormone therapy in patients with prostate and breast cancer),
21. Known hypersensitivity to any of the excipients of pembrolizumab, NB: L-histidine, L-Histidine Hydrochloride monohydrate, sucrose, polysorbate-80 (E433).

NB: L-histidine, L-Histidine Hydrochloride monohydrate, sucrose, polysorbate-80 (E433).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The rate of success of the experimental strategy at 6 months or after two successive colonoscopies (corresponding to timepoint at 6 months from the experimental strategy) following randomization. | 6 months
  The success at 6 months is defined as an absence of death, of disease progression, or of decision to perform surgery of the primary tumor for residual cells on biopsies, or for any other reason.

SECONDARY OUTCOMES:
The rate of strategy success at 24 months | 24 months
  The rate of strategy success at 24 months after randomization in the experimental arm
Incidence of Adverse Events (Safety assessment) | Up to 4 years
  Safety (according to NCI CTCAE v 5.0) of experimental strategy
Overall surival (OS) at 6, 12 and 24 months in both study arms | Up to 24 months
  OS is defined as the time between the date of randomization and the date of death from any cause. Survival data will be censored at the last follow-up.
Event-free survival (EFS) at 6, 12 and 24 months in both study arms | Up to 24 months
  EFS defined as the time from randomization to the first of the following events:
  * In experimental arm: death of all causes, PD, second primary CRC; decision to perform surgery of the primary tumor for residual cells on biopsies, or for any other reason.
  * In arm B: death of all causes, second primary CRC, local or metastatic relapse, whichever occurred first.
30-day and 90-day postoperative morbidity for patients who underwent surgery in both study arms | Up to 90 days post-surgery
  Postoperative morbidity is defined as a complication occurring during the hospital stay or within 30 or 90 days after surgery. Postoperative complications will be documented in a standardized form and their severity.
Time to deterioration (TTD) of health-related quality of life (HRQoL) | Up to 4 years
  TTD of HRQoL will be used to longitudinally analyze all HRQoL data (integrating all HRQoL measures). It is defined as the time interval between randomization in the study to the observation of a first deterioration of at least 10 points minimal clinically important difference (MCID) as compared to the baseline score. Meassurements at baseline, treatment visits, evaluation visits, end of treatment visit, and follow-up in both study arms.
Endoscopic complete response (ecR) assessment | Up to 24 months
  Endoscopy, accompanied by tissue biopsy, will be performed at months 3, 6, 9, 12, and 24 as a part of the watch-and-wait approach in the experimental arm. Endoscopy with biopsy of potential macroscopic lesions will be performed at 12 months in the arm B, as part of the standard of care.
  Endoscopic tumor response will be categorized as follows: clinical complete response (cCR), no visualization of tumor, white or red scar; nearly-cCR, minimal residual nodularity or stenosis; non-cCR, any ulcer with a necrotic bed regardless size, a definite residual mass, or nodularity. Clinical complete response is defined as the complete disappearance of the tumor and/or the absence of residual tumor cells on imaging, endoscopy, and biopsy.
Tumor regression grade (TRG) assessment | Up to 24 months
  TRG according to the Ryan score and the 8th American Joint Committee on Cancer tumor, node, metastasis (AJCC TNM) pathologic staging system in patients randomized in the experimental arm and who underwent surgery.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Institut Sainte Catherine, Avignon
  - CHU Besançon, Besançon
  - IHFB Cognacq Jay, Levallois-Perret
  - Centre Leon Berard, Lyon
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hôpital Saint Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Bordeaux Haut Lévêque, Pessac
  - CHU Poitiers, Poitiers
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No